CLINICAL TRIAL: NCT00520143
Title: Alglucosidase Alfa Temporary Access Program
Acronym: ATAP
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGLU03907
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Glycogen Storage Disease Type II (GSD-II); Pompe Disease (Late-Onset); Acid Maltase Deficiency Disease; Glycogenosis 2
Keywords: GSD-II, Pompe Disease, Glycogen Storage Disease II
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

INTERVENTIONS:
Biological: alglucosidase alfa (recombinant human acid alpha-glucosidase [rhGAA]) — IV infusion: 20mg/kg qow
  Other Names: Alglucosidase alfa

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The objective of this expanded access study is to provide patients with Pompe disease in the United States (US), access to alglucosidase alfa produced from a scaled up manufacturing process for a limited time until production at this scale is approved for commercial use by the Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* The patient or patient's legal guardian must provide signed, informed consent prior to performing any study-related procedures.
* The patient must reside in the US.
* The patient must have a confirmed diagnosis of Pompe disease defined as documented acid alpha-glucosidase (GAA) enzyme deficiency from any tissue source and/or GAA gene mutations.
* The patient must have/had documented clinical signs and symptoms of Pompe disease.
* The patient must have/had prior treatment with alglucosidase alfa produced at commercial scale OR be naive to enzyme replacement therapy (ERT) for the treatment of Pompe disease and meet at least 1 of the following criteria: require a wheelchair OR require some respiratory assistance for any number of hours (including night time) through non-invasive ventilation.
* The patient must be capable of complying with the required program schedule of assessments.

Exclusion Criteria:

* Females who are pregnant or lactating
* The patient has a clinical condition unrelated to Pompe disease that would interfere with program assessments.
* The patient is currently enrolled in any clinical studies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (74):
- United States (74):
  - Sheffield, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Prescott, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Bakersfield, California
  - Beverly Hills, California
  - Loma Linda, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Stanford, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Coral Springs, Florida
  - Daytona Beach, Florida
  - Gainsville, Florida
  - St. Petersburg, Florida
  - Decatur, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Augusta, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Lake Orion, Michigan
  - Rochester Hills, Michigan
  - Saint Joseph, Michigan
  - Minneapolis, Minnesota
  - Missoula, Montana
  - Omaha, Nebraska
  - Midland Park, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Corning, New York
  - Manhasset, New York
  - New York, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Jacksonville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Greenville, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - West Colombia, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Newport News, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
  - Pullman, Washington
  - Seattle, Washington
  - Morgantown, West Virginia
  - Green Bay, Wisconsin